CLINICAL TRIAL: NCT03421249
Title: Treatment of Knee Osteoarthrosis Using the Electromagnetic Fields: Blinded and Controlled Study
Brief Title: Treatment of Knee Osteoarthrosis Using the Electromagnetic Fields
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, Diego Galace de Freitas, Principal Investigator Diego Galace de Freitas, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hugo Cesar
Record Dates: First submitted 2018-01-08; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2016-01

CONDITIONS: Knee Osteoarthritis; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise; Magnetic Field Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A - Intervention (Active Comparator): Submitted to knee and hip muscle strengthening exercises and electromagnetic field therapy with Magnetron ® (Meditea - ARG) using the coplanar technique
  Interventions: Other: Exercises; Other: Electromagnetic field therapy
- Group B - exercises (Active Comparator): Performed exercises to strengthen the hip and knee muscles
  Interventions: Other: Exercises
- Group C - Placebo (Placebo Comparator): Performed hip and knee strengthening exercises and electromagnetic field therapy with the coplanar Magnetron® technique, but with the device switched off
  Interventions: Other: Electromagnetic field therapy
- Group D - Apparatus (Active Comparator): Only use electromagnetic field therapy with the coplanar Magnetron® technique
  Interventions: Other: Electromagnetic field therapy

INTERVENTIONS:
Other: Exercises — Muscle strengthening exercises of the hip and knee muscles
  Arms: Group A - Intervention; Group B - exercises
Other: Electromagnetic field therapy — Electromagnetic field therapy with Magnetron®
  Arms: Group A - Intervention; Group C - Placebo; Group D - Apparatus

SUMMARY:
This study is a randomized controlled clinical trial using a blind evaluator. Fifty-one volunteers were selected from 50 years to 70 years, obeying the following criteria: diagnosis of knee OA grade II and III through the radiographic classification of Kellgreen and Lawrence 1955, Body mass index (BMI) less than 40 kg / m², volunteers should have had knee pain for at least six months. All are from the Rehabilitation Sector of Santa Casa de Misericórdia de São Paulo (ISCMSP). The subjects were evaluated through a questionnaire developed by the authors of the study (Annex I), the Visual Analogue Scale (EVA) (Annex II), then applied to the Lower Extremity Functional Scale LEFS (Appendix III) and the Activities of daily living scale ADLs (Annex IV). In addition, the evaluation of muscular strength was through dynamometry using the Lafayete dynamometer model 01163, which was performed by a blind evaluator regarding the group that will belong to each candidate. The muscles tested were: quadriceps, ischiostibial and gluteus maximus. The randomization was through 60 brown envelopes divided into A, B, C and D, designating the randomness of the sample.

In addition to the initial evaluation, an evaluation was performed at the end of the tenth session and after 3 months of treatment.

The volunteers underwent a five-week treatment program, totaling 10 sessions, divided into four groups, group A - Intervention (INT) underwent knee and hip muscle strengthening exercises and electromagnetic field therapy with (Meditea - ARG) using the coplanar technique, group B - Exercises (EXE) carried out exercises to strengthen the hip and knee muscles in the C - Placebo group (PLA). hip and knee and electromagnetic field therapy with the Magnetron® coplanar technique, but with the device switched off and group D - Apparatus (APA) only use electromagnetic field therapy with the magnetron® coplanar technique. In the present study, there were no significant differences between groups regarding pain, function and muscle strength. However, group A obtained better results in the evaluated criteria, tending that the combination PEMF and exercises, is an indicated treatment for OA knee.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of knee OA grade II and III
* Body mass index (BMI) of less than 40 kg / m²
* knee pain for at least six months

Exclusion Criteria:

* Severe OA above grade 3
* previous physical therapy for at least 6 months,
* any other affection of the lower limbs (LLL) and lumbar spine,
* obesity (BMI> 40),
* patients with cardiovascular, metabolic, neurological, oncological or history of knee surgery.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Pain | The visual analog pain scale was performed without onset and after 3 months after treatment
  Visual Analog Pain Scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Added MAN, Added C, Kasawara KT, Rotta VP, de Freitas DG. Effects of a Knee Brace With a Patellar Hole Versus Without a Patellar Hole in Patients With Knee Osteoarthritis: A Double-Blind, Randomized Controlled Trial. Eval Health Prof. 2018 Dec;41(4):512-523. doi: 10.1177/0163278717714307. Epub 2017 Jun 30. PMID 28770628